CLINICAL TRIAL: NCT01175486
Title: The Effects of Thiazolidinedione on the Diabetic Retinopathy and Nephropathy
Brief Title: Thiazolidinedione (TZD) on the Diabetic Retinopathy and Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Tung-Ping Su, Chairman, Institutional Review Board, Taipei Veterans General Hospital,Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201004014IA
Record Dates: First submitted 2010-07-23; First posted 2010-08-04 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes
Keywords: thiazolidinediones; diabetes; retinopathy; nephropathy
MeSH Terms: conditions — Diabetes Mellitus; Retinal Diseases; Kidney Diseases | interventions — Pioglitazone; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Actos (Experimental): Actos 30 mg for 6 months
  Interventions: Drug: Actos (Pioglitazone)
- Acarbose (Active Comparator): Acarbose 50mg tid for 6 months
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Actos (Pioglitazone) — Actos 30 mg for 6 months
  Other Names: Pioglitazone
  Arms: Actos
Drug: Acarbose — Acarbose 50 mg tid for 6 months
  Other Names: Glucobay
  Arms: Acarbose

SUMMARY:
Objectives:

Thiazolidinediones (TZDs) are insulin sensitizers that decrease plasma glucose in type 2 diabetic patients. Thiazolidinediones can cause fluid retention and peripheral edema in diabetic patients, and the systematic fluid retention can be manifested as diabetic macular edema (DME). The overall goal of this study is to examine the effects of thiazolidinediones on the diabetic retinopathy and nephropathy.

Study design:

This is a prospective, randomized, open-labeled, controlled design to assess the effects thiozolidinediones on the diabetic retinopathy and nephropathy. The investigators will recruit 300 type 2 diabetic patients without significant retinopathy, nephropathy and cardiovascular disease. Inclusion criteria are type 2 diabetes, age between 30-80 years old, with microabluminuria, no significant retinopathy, on submaximal dose of sulphonylureas and metformin treatment, and A1C between 7-9%. Exclusion criteria are on insulin treatment, significant retinopathy and significant nephropathy. Patients with cardiovascular diseases, malignancy, pregnancy, in acute intercurrent illness, congestive heart failure, myocardial infarction, received PCI or CABG. All subjects will receive EKG and CXR before randomization.

These subjects will be randomized equally to 3 groups: acarbose, rosiglitazone and pioglitazone. The investigators will follow up for 6 months to investigate the short-term effects and 5 years to evaluate the long-term outcomes. The primary study end point of short-term study will be the macular thickness changes measured by optical coherence tomography, the changes in the level of urinary albumin-to-creatinine ratio, circulating metabolic parameters and adipocytokines during thiozolidinediones treatment. Secondary end point will be fasting blood glucose, A1C levels, development of clinically significant macular edema, serum creatinine change in patients with no history of diabetic retinopathy and nephropathy at baseline.

The primary study end point of long-term study will be the development of clinically significant macular edema and the time from the base-line visit to the first detection of overt nephropathy. Secondary end points include the development of greater than moderate NPDR, the time to the first event of the time from the base-line visit to a doubling of the serum creatinine concentration, end-stage renal disease, or death.

DETAILED DESCRIPTION:
The effects of thiazolidinedione on the diabetic retinopathy and nephropathy:

Overall Goal and Specific Aims

The overall goal of this study is to examine the effects of thiazolidinediones on the diabetic retinopathy and nephropathy.

The specific aims are:

1. To investigate the short-term effects of thiazolidinediones on the macular thickness measured by optical coherence tomography and the long-term effects of thiazolidinediones on the clinically significant macular edema and diabetic retinopathy documented by color photography and fluoroscein angiography.
2. Short-term effects of thiazolidinediones on the change of urine albumin excretion and serum cardiovascular risk profiles and long-term effects of thiazolidinediones on the estimated GFR change and progression to overt diabetic nephropathy.

Objectives

Thiazolidinediones (TZDs) are insulin sensitizers that decrease plasma glucose in type 2 diabetic patients. Thiazolidinediones can cause fluid retention and peripheral edema in diabetic patients, and the systematic fluid retention can be manifested as diabetic macular edema (DME). The overall goal of this study is to examine the effects of thiazolidinediones on the diabetic retinopathy and nephropathy.

Study design

This is a prospective, randomized, open-labeled, controlled design to assess the effects thiozolidinediones on the diabetic retinopathy and nephropathy. The investigators will recruit 300 type 2 diabetic patients without significant retinopathy, nephropathy and cardiovascular disease. Inclusion criteria are type 2 diabetes, age between 30-80 years old, with microabluminuria, no significant retinopathy, on submaximal dose of sulphonylureas and metformin treatment, and A1C between 7-9%. Exclusion criteria are on insulin treatment, significant retinopathy and significant nephropathy. Patients with cardiovascular diseases, malignancy, pregnancy, in acute intercurrent illness, congestive heart failure, myocardial infarction, received PCI or CABG. All subjects will receive EKG and CXR before randomization.

These subjects will be randomized equally to 3 groups: acarbose, rosiglitazone and pioglitazone. The investigators will follow up for 6 months to investigate the short-term effects and 5 years to evaluate the long-term outcomes. The primary study end point of short-term study will be the macular thickness changes measured by optical coherence tomography, the changes in the level of urinary albumin-to-creatinine ratio, circulating metabolic parameters and adipocytokines during thiozolidinediones treatment. Secondary end point will be fasting blood glucose, A1C levels, development of clinically significant macular edema, serum creatinine change in patients with no history of diabetic retinopathy and nephropathy at baseline.

The primary study end point of long-term study will be the development of clinically significant macular edema and the time from the base-line visit to the first detection of overt nephropathy. Secondary end points include the development of greater than moderate NPDR, the time to the first event of the time from the base-line visit to a doubling of the serum creatinine concentration, end-stage renal disease, or death.

The investigators also monitor the long-term safety issue, such as congestive heart failure, myocardial infarction, any cardiovascular event, and fracture.

Expected Results

TZDs can decrease plasma glucose in type 2 diabetic patients, but the major side effects are able to cause fluid retention. This prospective study will be able to test whether thiozolidinediones causes macular edema and to evaluate whether thiozolidinediones delays onset of diabetic retinopathy. The investigators also will be able to find the changes in the level of urinary albumin-to-creatinine ratio, circulating metabolic parameters and adipocytokines between the treatment of TZDs and Acrbose. The investigators can compare the time from the base-line visit to the first detection of overt nephropathy, the time to the first event of the composite end point of the time from the base-line visit to a doubling of the serum creatinine concentration, end-stage renal disease, or death.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age between 30-80 years old
* No significant nephropathy
* No significant retinopathy
* On submaximal dose of sulphonylureas and metformin treatment
* A1C between 7-9%

Exclusion Criteria:

* On insulin treatment
* Significant retinopathy (greater than moderate non-proliferative retinopathy)
* Significant nephropathy (overt proteinuria or serum Cr >1.50 mg/dL)
* Malignancy
* Pregnancy
* Acute intercurrent illness
* Congestive heart failure (CHF, according to New York heart Association, NYHA functional class III to IV)
* Myocardial infarction, received PCI or CABG or liver cirrhosis

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Diabetic retinopathy | 6 months
  The macular thickness changes
Diabetic nephropathy | 6 months
  The changes in the level of urinary albumin-to-creatinine ratio

SECONDARY OUTCOMES:
Diabetic retinopathy | 3 years
  Development of greater than moderate NPDR, clinically significant macular edema
Diabetic nephropathy | 3 years
  The change of urine albumin excretion, estimated GFR change, progression to overt diabetic nephropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Harn-Shen Chen, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taiwan, Taipei, Taiwan

REFERENCES:
- [Derived] Chen YH, Tarng DC, Chen HS. Renal Outcomes of Pioglitazone Compared with Acarbose in Diabetic Patients: A Randomized Controlled Study. PLoS One. 2016 Nov 3;11(11):e0165750. doi: 10.1371/journal.pone.0165750. eCollection 2016. PMID 27812149